CLINICAL TRIAL: NCT04747301
Title: The Effectiveness and Safety of Double-balloon Versus Vaginal Prostaglandin for Cervical Ripening in Women With Low-risk Pregnancies: A Randomized Controlled Trial (DOBA-PRO)
Brief Title: DOuble-BAlloon Versus PROstaglandin E2 for Cervical Ripening in Low Risk Pregnancies
Acronym: DOBA-PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Obstetrics and Gynecology Hospital (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSHN.0001.2021
Record Dates: First submitted 2021-01-22; First posted 2021-02-10 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Induction of Labor
Keywords: Induction of labor; Low-risk pregnancies; Double-balloon catheter; Prostaglandin E2
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Intervention Model Description: Low-risk pregnant women eligible for study will be asked to sign the informed consent form. Then, they will be randomly assigned in a 1:1 ratio to receive either double balloon insertion or vaginal prostaglandin E2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-balloon catheter group (Other): Sweeping the membranes by UTAH CVX-RIPE® (Utah Medical Products, Inc, 7043 South 300 West, Midvale, Utah 84047 USA).
  Interventions: Device: Double-balloon catheter (UTAH CVX-RIPE) for cervical ripening
- Vaginal insertion Prostaglandin E2 group (Other): Propess® 10mg Vaginal delivery system (Ferring Controlled Therapeutics Ltd., 1 Redwood Place, Peel Park Campus, East Kilbride, Glasgow, G74 5PB, UK) is a vaginal insert containing 10mg of dinoprostone in a timed-release formulation (the medication is released at 0.3 mg/hour).
  Interventions: Drug: Dinoprostone 10mg (Propess)

INTERVENTIONS:
Device: Double-balloon catheter (UTAH CVX-RIPE) for cervical ripening — Sweeping the membranes by UTAH CVX-RIPE® (Utah Medical Products, Inc, 7043 South 300 West, Midvale, Utah 84047 USA). The catheter will be inserted manually until the proximal balloon is in the cervical canal, the distal balloon should be intrauterine and in the extra-amniotic space. The intrauterine balloon is inflated with 40mL saline and retracted so that it rests against the internal oz. The proximal balloon should now be outside the external oz and is inflated with 20mL saline. If the balloons are correctly situated on both ends of the cervix, they can be inflated with up to 80mL saline each.
  Cardiotocograph will be performed 30min, 2 hours after insertion and every 6 hours. The balloon is placed for a maximum of 24 hours.
  If it is expelled in the first 12 hours and the patient has no contractions or still shows an unfavorable cervix, another balloon is placed for a maximum of another 24 hours.
  The patients will be examined in case of extremely painful or membranes ruptured.
  Arms: Double-balloon catheter group
Drug: Dinoprostone 10mg (Propess) — Propess® 10mg Vaginal delivery system (Ferring Controlled Therapeutics Ltd., 1 Redwood Place, Peel Park Campus, East Kilbride, Glasgow, G74 5PB, UK) is a vaginal insert containing 10mg of dinoprostone in a timed-release formulation (the medication is released at 0.3 mg/hour).
  A Propess vaginal system is inserted by a research doctors. As in the catheter procedure, Fetal Heart Rate is monitored 30min before and 2 hours after placement. Cardiotocograph and vaginal examination will be performed every 6 hours. The vaginal system is placed for a maximum of 24 hours.
  If it is expelled in the first 12 hours and the patient has no contractions or still shows an unfavorable cervix, another vaginal system is placed for a maximum of another 24 hours.
  The patients will be examined in case of extreme pain or membranes ruptured.
  Other Names: Vaginal Prostaglandin E2 (Propess)
  Arms: Vaginal insertion Prostaglandin E2 group

SUMMARY:
To compare the effectiveness and safety of double balloon catheter and vaginal insert Prostaglandin E2 in cervical ripening prior to Induction of Labor in low-risk women from 39+0 to 40+6 weeks of gestation.

DETAILED DESCRIPTION:
Induction of labor (IOL) is a technique to establish vaginal delivery when the risks for continuing the pregnancy for mother or baby are higher than the risks of delivery. In case the cervix is unripe, cervical ripening before the onset of labor is needed. The two main mechanisms of cervical ripening can be categorized as mechanical or pharmacological.

A Cochrane systematic review and other recent meta-analysis have shown that cervical ripening with a balloon is probably as effective as induction of labor with vaginal Prostaglandin E2. However, this conclusion is based on low to moderate quality evidence. Only a limited number of randomized clinical trials (RCTs) have been conducted. Many of those suffering from small sample sizes and different study subjects, i.e. high-risk subjects only, and mixed population.

In current practice, induction of labor is not only used in high-risk patients with clear indications for pregnancy termination. The ARRIVE trial has shown a significant benefit of labor induction over expectant management among the low-risk population. Based on this evidence, the American College of Obstetricians and Gynecologists (ACOG) has suggested: "It's time to induce of labor at 39th week of gestation". Since then, there is a trend in favoring elective induction before the due date over expectant management. Besides, more and more pregnant women want to shorten the duration of pregnancy or to time the birth of the baby due to the convenience of the mother and/or healthcare workers.

This makes the optimal method of Induction of Labor in terms of effectiveness and safety for both mothers and their babies even more important. In this study, the investigators will compare the effectiveness and safety of double-balloon catheter and Prostaglandin E2 for elective labor induction in low-risk pregnancies.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age ≥ 18
2. Singleton pregnancy. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks gestational age.
3. Gestational age at randomization from at 39+0 to 40+6 weeks of gestation.
4. Cephalic presentation
5. Intact membrane
6. Unfavourable cervix (Bishop<6)
7. Informed consent

Exclusion Criteria:

1. Maternal medical illness associated with increased risk of adverse pregnancy outcome (any diabetes mellitus, any hypertensive disorders, cardiac diseases, renal insufficiency, systemic lupus erythematosus, mental disorders, HIV positive, use of heparin or low-molecular weight heparin during the current pregnancy etc.)
2. Abnormal placenta: Active vaginal bleeding greater than bloody show or placenta previa, accreta or vasa previa
3. Abnormal amniotic fluid volume:

   * Oligohydramnios (MVP < 2cm)
   * Polyhydramnios (MVP > 10cm)
4. Abnormal fetus

   * Fetal demise or known major fetal anomalies
   * Fetal growth restriction (FGR) (EFW < 3% or < 10% and abnormal Doppler)
   * Non-reassuring fetal status (no fetal movements, abnormal fetal heart rate at auscultation)
5. Previous C-section
6. Planned for C-section or contra-indication to labour
7. Cerclage or use of pessary in current pregnancy
8. Refusal of blood product.
9. Participation in another interventional study that influences management of labour at delivery or perinatal morbidity or mortality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants delivered vaginally | From randomization until delivery, assessed up to 3 days after randomization
  Number of participants delivered vaginally

SECONDARY OUTCOMES:
Number of participants with Side - effect of induction's method | From induction until delivery, assessed up to 3 days after induction
  Including any of: nausea, vomiting, diarrhea, pain...
Number of participants using more than one induction agent required | From induction until delivery, assessed up to 3 days after induction
  Number of participants using more than one induction agent required
Number of participants having oxytocin augmentation | From induction until delivery, assessed up to 3 days after induction
  Number of participants having oxytocin augmentation
Number of participants with uterine tachysystole | From induction until delivery, assessed up to 3 days after induction
  Defined as more than 5 contractions in 10 minutes over a minimal period of two times 10 minutes with Fetal Heart Rate changes and/or a contraction lasting more than 3 minutes with Fetal Heart Rate changes.
Time from induction of labor to delivery | From induction until delivery, assessed up to 3 days after induction
  Duration from induction to delivery (hours)
Number of participants delivered vaginally within 24 hours | Within 24 hours from labor induction
  Number of participants delivered vaginally within 24 hours
Number of participants with post-partum haemorrhage | Within 24 hours from delivery
  Defined as blood loss >500 ml at vaginal birth or >1000 ml at caesarean birth within 24 hours after birth
Number of participants having uterine atony | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Use of two or more uterotonics other than oxytocin; other surgical interventions such as uterine compression by hands and/or sutures, uterine artery ligation, embolization, hypogastric ligation, or balloon tamponade).
Number of participants having maternal post-partum blood transfusion | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants having maternal post-partum blood transfusion
Number of participants with hypertension complications | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants with hypertension complications
Number of participants with uterine dehiscence or rupture | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Uterine dehiscence (defined as clinically asymptomatic disruption of the uterus that is discovered incidentally at surgery) or rupture (defined as clinically significant rupture involving the full thickness of the uterine wall and requiring surgical repair)
Number of participants with maternal infection | From induction until maternal hospital discharge, assessed up to 28 days after induction
  * Fever (defined as a temperature ≥37.5 degrees Celsius)
  * Start of intravenous broad-spectrum antibiotics (with evidence of infection confirmed by clinical and subclinical presentation)
  * Endometritis, myometritis or urinary tract infection (proven positive vaginal discharge/urine culture)
Number of participants with hysterectomy | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Hysterectomy for any postpartum complications
Number of participants with damage to internal organs | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Including intestines, bladder or ureters
Number of participants with other post-partum complications | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Includes: venous embolism, pulmonary embolism, stroke, cardiac arrest
Number of participants admitted to intensive care unit | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants admitted to intensive care unit
Number of maternal death among participants | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Maternal death from randomization through hospital discharge
Number of participants referred to other hospital due to severe morbidities | From randomization until maternal hospital referral, assessed up to 28 days after randomization
  Including: pulmonary embolus, stroke, cardiorespiratory arrest, etc.
Maternal length of stay | From admission until maternal hospital discharge, assessed up to 28 days after admission
  Duration of stay in hospital (days)
Psychometric aspects | At admission (version A) and before maternal hospital discharge (version B), assessed up to 28 days after admission
  Feelings and thoughts pregnant women at antepartum and postpartum will be evaluated by Wijma Delivery Expectancy/Experience Questionnaires' (W-DEQ) version A and version B, respectively, expected to be filled out in approximately 30 minutes
  This is a questionnaire which measures a construct of fear related to childbirth during pregnancy and after delivery by asking the woman about her expectancies before delivery(version A) - performed at admission, and experiences after delivery (version B) - performed before maternal hospital discharge respectively.
  When filling in the W-DEQ, the woman is instructed to rate her personal feelings and cognitions on a six-point scale. The minimum score is 0 and the maximum score is 126. The higher the score, the greater the fear of childbirth manifested.
Apgar scores at 1 and 5 minute | Assessed at 1 and 5 minute after birth
  Apgar scores at 1 and 5 minute
Number of Infants with Apgar Score ≤7 at 1 and 5 minutes | Assessed at 1 and 5 minute after birth
  Infants with Apgar Score ≤7 at 1 and 5 minutes
Number of neonates admitted to the Neonatal Intensive Care Unit or Intermediate care unit | From delivery until admission to Neonatal Intensive Care Unit or Intermediate care unit, assessed up to 7 days after delivery
  Number of neonates admitted to the Neonatal Intensive Care Unit or Intermediate care unit
Reason for Neonatal Intensive Care Unit admission | From delivery until Neonatal Intensive Care Unit admission, assessed up to 28 days after delivery
  Reason for Neonatal Intensive Care Unit admission such as: respiratory distress, hypoglycemia, seizures, etc.
Length of stay at the Neonatal Intensive Care Unit or Intermediate care unit | From admission to Neonatal Intensive Care Unit/ Intermediate care unit until neonatal discharge or hospital referral, assessed up to 28 days after Neonatal Intensive Care Unit admission
  Duration from admission to Neonatal Intensive Care Unit or Intermediate care unit to Neonatal Intensive Care Unit/ Intermediate care unit discharge or hospital referral
Number of neonates with birth trauma | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Include: bone fractures, traumatic pneumothorax, facial nerve palsy, other neurologic injury (Brachial plexus palsy...), etc.
Number of neonates with hypoglycemia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with hypoglycemia
Number of neonates with jaundice and hyperbilirubinemia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with jaundice and hyperbilirubinemia
Number of neonates with Hypoxic ischemic encephalopathy or need for therapeutic hypothermia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with Hypoxic ischemic encephalopathy or need for therapeutic hypothermia
Number of neonates with meconium aspiration syndrome | From delivery until neonatal hospital discharge, assessed up to 07 days after delivery
  Criteria include:
  * Meconium-stained amniotic fluid
  * Respiratory distress at birth or shortly after birth
  * Characteristic radiographic features: The initial chest film may show streaky, linear densities -> the lungs typically appear hyper-inflated with flattening of the diaphragms.
Number of neonates in need for respiratory supports | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Incubation, Continuous Positive Airway Pressure, or high-flow nasal cannula (HFNC) for ventilation or cardiopulmonary resuscitation within the first 72 hours
Number of neonates with neonatal infection | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid (CSF), or catheterized/supra-pubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an X-ray confirming infection
Number of neonates with neonatal seizures | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with neonatal seizures
Number of neonates with intracranial hemorrhage | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Intra-ventricular hemorrhage grades III and IV, subgaleal hematoma, subdural hematoma, or subarachnoid hematoma Subgaleal hematoma, subdural hematoma, or subarachnoid hematoma
Number of neonates need blood transfusion | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates need blood transfusion
Number of neonatal deaths | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Includes: Intrapartum/neonatal/perinatal deaths
Number of neonates referred to other hospital for severe morbidities | From delivery until neonatal hospital referral, assessed up to 28 days after delivery
  Number of neonates referred to other hospital for severe morbidities

CONTACTS AND LOCATIONS:
Overall Officials: Ben W Mol, PhD. MD, Study Chair — Monash University; Anh Nguyen Duy, PhD. MD, Study Director — Hanoi Obstetric and Gynecology Hospital; Vinh Dang Quang, PhD. MD, Principal Investigator — Mỹ Đức Hospital; Ha Nguyen Thi Thu, PhD. MD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital
Locations (1):
- Hanoi Obstetrics and Gynecology Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du YM, Zhu LY, Cui LN, Jin BH, Ou JL. Double-balloon catheter versus prostaglandin E2 for cervical ripening and labour induction: a systematic review and meta-analysis of randomised controlled trials. BJOG. 2017 May;124(6):891-899. doi: 10.1111/1471-0528.14256. Epub 2016 Aug 17. PMID 27533177
- [Background] Liu YR, Pu CX, Wang XY, Wang XY. Double-balloon catheter versus dinoprostone insert for labour induction: a meta-analysis. Arch Gynecol Obstet. 2019 Jan;299(1):7-12. doi: 10.1007/s00404-018-4929-8. Epub 2018 Oct 12. PMID 30315411
- [Background] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2019 Oct 18;10(10):CD001233. doi: 10.1002/14651858.CD001233.pub3. PMID 31623014
- [Background] Shechter-Maor G, Haran G, Sadeh-Mestechkin D, Ganor-Paz Y, Fejgin MD, Biron-Shental T. Intra-vaginal prostaglandin E2 versus double-balloon catheter for labor induction in term oligohydramnios. J Perinatol. 2015 Feb;35(2):95-8. doi: 10.1038/jp.2014.173. Epub 2014 Oct 2. PMID 25275693
- [Background] Du C, Liu Y, Liu Y, Ding H, Zhang R, Tan J. Double-balloon catheter vs. dinoprostone vaginal insert for induction of labor with an unfavorable cervix. Arch Gynecol Obstet. 2015 Jun;291(6):1221-7. doi: 10.1007/s00404-014-3547-3. Epub 2014 Nov 19. PMID 25408273
- [Background] Wang W, Zheng J, Fu J, Zhang X, Ma Q, Yu S, Li M, Hou L. Which is the safer method of labor induction for oligohydramnios women? Transcervical double balloon catheter or dinoprostone vaginal insert. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1805-8. doi: 10.3109/14767058.2014.880880. Epub 2014 Feb 3. PMID 24397441
- [Background] Cromi A, Ghezzi F, Uccella S, Agosti M, Serati M, Marchitelli G, Bolis P. A randomized trial of preinduction cervical ripening: dinoprostone vaginal insert versus double-balloon catheter. Am J Obstet Gynecol. 2012 Aug;207(2):125.e1-7. doi: 10.1016/j.ajog.2012.05.020. Epub 2012 Jun 1. PMID 22704766
- [Background] Suffecool K, Rosenn BM, Kam S, Mushi J, Foroutan J, Herrera K. Labor induction in nulliparous women with an unfavorable cervix: double balloon catheter versus dinoprostone. J Perinat Med. 2014 Mar;42(2):213-8. doi: 10.1515/jpm-2013-0152. PMID 24096438
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Dos Santos F, Drymiotou S, Antequera Martin A, Mol BW, Gale C, Devane D, Van't Hooft J, Johnson MJ, Hogg M, Thangaratinam S. Development of a core outcome set for trials on induction of labour: an international multistakeholder Delphi study. BJOG. 2018 Dec;125(13):1673-1680. doi: 10.1111/1471-0528.15397. Epub 2018 Sep 10. PMID 29981523